CLINICAL TRIAL: NCT07057791
Title: Phase II Dose Optimization Study of Platinum/Etoposide Plus Ivonescimab (CEI) as First-Line Treatment of Extensive-Stage Small Cell Lung Cancer
Brief Title: Phase II Study of Platinum/Etoposide Plus Ivonescimab for Extensive-Stage Small Cell Lung Cancer
Acronym: PrE0510
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: PrECOG, LLC. (Other)
Collaborators: Summit Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PrE0510
Record Dates: First submitted 2025-06-30; First posted 2025-07-10 (Actual); Last update posted 2026-01-27 (Actual); Status verified 2026-01

CONDITIONS: Extensive Stage Lung Small Cell Cancer
Keywords: Extensive Stage Small Cell Lung Cancer; Small Cell Lung Cancer; Ivonescimab; Carboplatin; Etoposide
MeSH Terms: conditions — Small Cell Lung Carcinoma

STUDY DESIGN:
Intervention Model Description: Open label, randomized (1:1) trial of ivonescimab 10 mg/kg versus 20 mg/kg with carboplatin and etoposide during induction followed by ivonescimab (at dose received during induction) until progression. Participants will be stratified by Eastern Cooperative Oncology Group (ECOG) Performance Status (0/1) and Brain Metastases (Yes/No).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Arm A: Ivonescimab 10 mg/kg (Experimental): Induction with ivonescimab 10 mg/kg, carboplatin and etoposide every 21 days x 4 cycles followed by maintenance ivonescimab 10 mg/kg every 21 days until progression, unacceptable toxicity or participant withdrawal. Up to 24 months of ivonescimab from cycle 1 day 1 of Induction.
  Interventions: Drug: Ivonescimab 10 mg/kg
- Arm B: Ivonescimab 20 mg/kg (Experimental): Induction with ivonescimab 20 mg/kg, carboplatin and etoposide every 21 days x 4 cycles followed by maintenance ivonescimab 20 mg/kg every 21 days until progression, unacceptable toxicity or participant withdrawal. Up to 24 months of ivonescimab from cycle 1 day 1 of Induction.
  Interventions: Drug: Ivonescimab 20 mg/kg

INTERVENTIONS:
Drug: Ivonescimab 10 mg/kg — Induction every 21 days x 4 cycles: Ivonescimab 10 mg/kg intravenous (IV) on Day 1 followed by carboplatin area under the curve (AUC) 5 IV on Day 1 and etoposide 100 milligrams per square meter (mg/m²) IV on Day 1, 2 and 3 followed by maintenance ivonescimab 10 mg/kg every 21 days until progression, unacceptable toxicity or participant withdrawal. Up to 24 months of ivonescimab from cycle 1 day 1 of Induction.
  Other Names: AK112; SMT112; Akeso
  Arms: Arm A: Ivonescimab 10 mg/kg
Drug: Ivonescimab 20 mg/kg — Induction every 21 days x 4 cycles: Ivonescimab 20 mg/kg IV on Day 1 followed by carboplatin AUC 5 IV on Day 1 and etoposide 100 mg/m² IV on Day 1, 2 and 3 followed by maintenance ivonescimab 20 mg/kg every 21 days until progression, unacceptable toxicity or participant withdrawal. Up to 24 months of ivonescimab from cycle 1 day 1 of Induction.
  Other Names: AK112; SMT112; Akeso
  Arms: Arm B: Ivonescimab 20 mg/kg

SUMMARY:
Eligible untreated participants with Extensive Stage Small Cell Lung Cancer (ES-SCLC) who are ≥ 18 years of age will be randomized to receive ivonescimab 10 milligrams per kilogram (mg/kg) or ivonescimab 20 mg/kg in combination with carboplatin and etoposide.

Ivonescimab is a type of drug called a bispecific antibody. Antibodies are proteins that specifically recognize and bind to other types of proteins called antigens. Antibodies and antigens can work together to help the immune system fight cancer cells. Bispecific antibody, meaning it targets two different molecules at the same time.

Ivonescimab is a new drug that may help the immune system attack cancer cells and may also block certain pathways that cancer uses to grow and spread. This dual action of ivonescimab aims to help the immune system to fight the cancer and also disrupt tumor growth by blocking blood vessel formation that tumors use to grow.

Participants will receive induction with 4 cycles of ivonescimab (dose determined by randomization) with standard of care carboplatin and etoposide followed by maintenance therapy with ivonescimab at the same dose received during induction. Treatment will continue until disease progression, unacceptable toxicity or participant withdrawal.

The purpose of this study is to determine what dose of ivonescimab works best in combination with carboplatin and etoposide chemotherapy in ES-SCLC. We will also examine the side effects, good and bad, associated with ivonescimab.

DETAILED DESCRIPTION:
Randomized, Phase II, open-label trial designed to determine the optimal dose of ivonescimab with carboplatin and etoposide for a more diverse Western participant population with ES- SCLC based on overall response rate and safety profile of two dose levels of ivonescimab (10 mg/kg versus 20 mg/kg) previously evaluated in the Chinese population.

The simultaneous blockade of vascular endothelial growth factor (VEGF) and Programmed Death-Ligand 1 (PDL-1) by ivonescimab may achieve a higher target binding of VEGF and PD-1 within the tumor microenvironment and produce increased anti-tumor effect with an improved safety profile than administration of anti-PD-(L)1 and anti-VEGF therapies separately.

Participants will be randomized 1:1 to receive ivonescimab 10 mg/kg or 20 mg/kg. Induction treatment will be administered on a 21-day cycle for four cycles with standard of care carboplatin and etoposide.

Following the induction phase, participants will continue maintenance therapy with ivonescimab on a 21-day cycle at the dose received during induction (10 mg/kg or 20 mg/kg). Treatment will be discontinued in all participants who have evidence of progressive disease by Response Criteria Evaluation in Solid Tumors version 1.1 (RECIST v1.1).

Research tumor tissue will be requested at baseline for future research. Research blood samples will also be obtained for future research which may include measuring the level of ivonescimab in the blood and immune responses or antibodies to ivonescimab.

ELIGIBILITY:
Selection Criteria:

* Patients must have pathologically confirmed Extensive Stage Small Cell Lung Cancer (ES-SCLC).
* No prior systemic therapy for the disease under study (ES-SCLC).
* Patients must have measurable disease according to Response Evaluation Criteria for Solid Tumors (RECIST) v1.1.
* Patient must be ≥ 18 years of age.
* Patient must have an ECOG performance status of 0-1.
* Patient must have the ability to understand and willingness to sign a written informed consent document.
* Willing to provide archived tumor tissue (if sufficient tumor tissue available) and blood samples for research.
* Patient must have adequate organ function and marrow function as defined below, obtained ≤ 14 days prior to registration/randomization. No blood transfusions or growth factor therapy allowed within 7 days of screening labs.

  * Absolute Neutrophil Count (ANC) ≥ 1500/microliter (mcL)
  * Platelets ˃100,000/mcL
  * Hemoglobin >9.0 gram/deciliter (g/dL)
  * Prothrombin time (PT) or international normalized ratio (INR) ≤ 1.5x Upper Limit Normal (ULN), and partial prothrombin time (PTT) or activated partial thromboplastin time (aPTT) ≤ 1.5x ULN
  * Serum Creatinine ≤ 2x ULN
  * Creatinine clearance (CrCl) ≥ 50 milliliter/minute (mL/min)
  * Urine Protein <2+
  * Alanine Aminotransferase (ALT) and Aspartate Aminotransferase (AST) ≤ 2.5x ULN or ≤ 5x ULN for patients with liver metastasis
  * Total Bilirubin ≤ 1.5x ULN or ≤ 3x ULN for patients with liver metastasis or suspected/documented Gilbert's disease
* Patient must not be pregnant or breast-feeding due to the potential harm to an unborn fetus and possible risk for adverse events in nursing infants with the treatment regimens being used.
* Patient must not expect to conceive or father children by using an accepted and effective method(s) of contraception or by abstaining from sexual intercourse for the duration of their participation in the study, and for 120 days after the last dose of study drug(s).
* Patients must not have symptomatic central nervous system (CNS) metastases, CNS metastasis ≥ 1.5 cm, CNS radiation within 7 days prior to randomization, potential need for CNS radiation within the first cycle, or leptomeningeal disease.
* Patients must not have imaging during the screening period that shows:

  1. Radiologically documented evidence of major blood vessel invasion (central pulmonary artery, central pulmonary veins, aorta, brachiocephalic artery, common carotid artery, subclavian artery, superior vena cava) or tumor invading organs (heart, trachea, esophagus, central bronchi [not including segmental bronchi]) or if there is a risk of esophagotracheal or esophagopleural fistula .
  2. Radiographic evidence of major blood vessel encasement with narrowing of the vessel or intratumor lung cavitation or necrosis that the investigator determines will pose a significantly increased risk of bleeding.
* Patients with a prior or concurrent malignancy whose natural history or treatment does not have the potential to interfere with the safety or efficacy assessment of the investigational regimen are eligible for this trial.
* Patients must not have major surgical procedures or serious trauma within 28 days prior to randomization or plans for major surgical procedures within 28 days after the first dose.
* Patients must not have history of bleeding tendencies or coagulopathy and/or clinically significant bleeding symptoms or risk within 4 weeks prior to randomization, including but not limited to:

  1. Hemoptysis (defined as coughing up ≥ 0.5 teaspoon of fresh blood or small blood clots). Transient hemoptysis associated with diagnostic bronchoscopy is allowed.
  2. Nasal bleeding/epistaxis (bloody nasal discharge is allowed).
  3. Current use of prophylactic or full-dose anticoagulants or anti-platelet agents for therapeutic purposes that is not stable prior to randomization is not allowed.
* Patients must not have history of major diseases before randomization, specifically:

  1. Unstable angina, myocardial infarction, congestive heart failure (New York Heart Association (NYHA) classification ≥ Grade 2) or unstable vascular disease (e.g., aortic aneurysm at risk of rupture, Moyamoya disease) that required hospitalization within 12 months prior to randomization, or other cardiac impairment that may affect the safety evaluation of the study drug (e.g., poorly controlled arrhythmias, myocardial ischemia).
  2. History of any grade arterial thromboembolic event, Grade 3 and above venous thromboembolic event, as specified in National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) 5.0, transient ischemic attack, cerebrovascular accident, hypertensive crisis, or hypertensive encephalopathy within 12 months prior to randomization.
  3. History of esophageal gastric varices, severe ulcers, wounds that do not heal, abdominal fistula, intra-abdominal abscesses, or acute gastrointestinal bleeding within 6 months prior to randomization.
  4. History of perforation of the gastrointestinal tract and/or fistula, history of gastrointestinal obstruction (including incomplete intestinal obstruction requiring parenteral nutrition), extensive bowel resection (partial colectomy or extensive small bowel resection) within 6 months prior to randomization.
* Patients must not have poorly controlled hypertension with repeated systolic blood pressure ≥ 150 mmHg or diastolic blood pressure ≥ 100 mmHg after oral antihypertensive therapy.
* Patients must not have prolongation of QTc interval >480 msec
* Patients must not have active autoimmune or lung disease requiring systemic therapy (e.g., with disease modifying drugs, prednisone >10 mg daily or equivalent, immunosuppressant therapy) within 2 years prior to randomization.
* Patients must not have severe infection within 4 weeks prior to randomization, including but not limited to comorbidities requiring hospitalization, sepsis, or severe pneumonia; active infection requiring systemic anti-infective therapy within 2 weeks prior to randomization (excluding antiviral therapy for hepatitis B or C).
* Patients must not have uncontrolled pleural effusions, pericardial effusions, or ascites that is clinically symptomatic.
* Patients must not have history of non-infectious pneumonia requiring systemic corticosteroids, or current interstitial lung disease.
* Patients must not have active or prior history of inflammatory bowel disease (e.g., Crohn's disease, ulcerative colitis, or chronic diarrhea.
* Patients must not have pre-existing peripheral neuropathy ≥ Grade 2 by CTCAE V5.0.
* Human immunodeficiency virus (HIV)-infected patients on effective anti-retroviral therapy with undetectable viral load within 6 months of registration/randomization are eligible for this trial.
* Patient must not have received any live vaccine within 28 days prior to registration/randomization.
* Patients with a known allergy to any of the study medications, their analogues, or excipients in the various formulations of any agent are not eligible.
* Patients with any serious medical or psychiatric illness that could, in the investigator's opinion, potentially interfere with the completion of the treatment according to the protocol are not eligible.
* Patients may not participate in any other therapeutic clinical trials, including those with other investigational agents not included in this trial during treatment on this study without prior approval from PrECOG.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2026-02 (Estimated); Primary Completion 2027-12 (Estimated); Study Completion 2030-01 (Estimated)

PRIMARY OUTCOMES:
Optimal Dose of Ivonescimab in Combination with Carboplatin and Etoposide - Overall Response Rate (ORR) | 18 months
  Overall Response Rate (ORR) defined as the proportion of participants achieving complete response (CR) or partial response (PR) as best response on treatment based on RECIST v1.1 criteria at each dose level.
Optimal Dose of Ivonescimab in Combination with Carboplatin and Etoposide - Grade 3-5 Treatment-Related Toxicity Rate | 18 months
  All grade 3-5 adverse events (AE) with treatment attribution of possibly, probably or definite based on Common Terminology Criteria for Adverse Events Version 5.0 (CTCAE V5.0) that are not resolved in accordance with treatment guidelines will be counted. Rate is the proportion of treated participants experiencing at least one of these adverse events as defined during the time of observation.

SECONDARY OUTCOMES:
Progression-Free Survival (PFS) of Ivonescimab in Combination with Carboplatin and Etoposide | 18 months
  PFS based on the Kaplan-Meier method defined as the duration between randomization and documented disease progression (PD) defined per RECIST 1.1 criteria. or death, or is censored at time of last disease assessment.
Overall Survival (OS) of of Ivonescimab in Combination with Carboplatin and Etoposide | 24 months
  OS based on the Kaplan-Meier method defined as the time from study entry to death or censored at date last known alive.
Disease Control Rate (DCR) of Ivonescimab in Combination with Carboplatin and Etoposide | 18 months
  DCR defined as the proportion of participants who achieved a best overall response of complete response (CR), partial response (PR) , or stable disease (SD), as determined by investigator assessment (disease control rate- CR+PR+SD) per RECIST v1.1. Patients who have not progressed by the time of analysis will be censored at the date they are last known to be alive and progression-free.
Duration of Response (DoR) of Ivonescimab in Combination with Carboplatin and Etoposide | 18 months
  DoR is defined as from the time measurement criteria are first met for CR/PR (whichever is first recorded) until the first date that recurrent or progressive disease is objectively documented. Patients who have not progressed by the time of analysis will be censored at the date they are last known to be alive and progression-free.
Duration of Stable Disease of Ivonescimab in Combination with Carboplatin and Etoposide | 18 months
  Duration of stable disease is measured from the start of treatment until the criteria for disease progression are met per RECIST v1.1. Patients who have not progressed by the time of analysis will be censored at the date they are last known to be alive and progression-free.

CONTACTS AND LOCATIONS:
Overall Officials: Taofeek Owonikoko, MD, PhD, Study Chair — University of Maryland, Baltimore
Locations (1):
- Aspirus Cancer Center Wausau, Wausau, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: No
Data is proprietary.